CLINICAL TRIAL: NCT05623462
Title: Virtual Reality Treadmill Training for Improving Gait Performance in the Elderly
Brief Title: Virtual Reality Training for Walking Improvement in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umm Al-Qura University (Other)
Responsible Party: Principal Investigator, Ehab Mohamed Abd El Kafy, Professor of Physical Therapy, Umm Al-Qura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22UQU428521DSR01
Record Dates: First submitted 2022-11-11; First posted 2022-11-21 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2022-11

CONDITIONS: Gait, Unsteady
Keywords: Gait; Older Adults; Virtual Reality
MeSH Terms: conditions — Gait Disorders, Neurologic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Active Comparator): Participants in the control group will receive conventional gait training (conventional physical therapy program) for one hour as the following.
  * Part (1) Treadmill gait training without virtual reality. (for 30 minutes)
  * Rest for 15 minutes between the first part and the second part.
  * Part (2) Indoor open environment gait training exercises(over-ground gait training exercises.). (for 30 minutes)
  Interventions: Other: Conventional Physical Therapy Program
- Experimental Group (Experimental): Participants in the experimental group will receive a treatment program that is comprised of two parts.
  * The first part included training, for (30 minutes), on The C-Mill virtual reality treadmill. The C-Mill is an instrumented treadmill with interactive virtual reality games and applications. The C-Mill applies an augmented virtual reality environment, obstacle avoidance games, and a variety of balance challenges in a safe and controlled environment to increase walking adaptability and performance in everyday life.
  * There will be 15 minutes rest between parts one and two of the training program
  * The second part (conventional training program) (30 minutes) will include: Indoor open environment gait training exercises (over-ground gait training exercises.). (30 minutes)
  Interventions: Device: The C-Mill virtual reality treadmill

INTERVENTIONS:
Device: The C-Mill virtual reality treadmill — The C-Mill treadmill is an innovative device used for the training of impaired gait and balance. The C-Mill is an instrumented treadmill with interactive virtual reality games and applications.The instrument is supplied with a safety frame, body weight support, treadmill force plates, treadmill belt, adjustable handrails, cameras, user operating system, interactive visual screen and augmented reality projection.
  Arms: Experimental Group
Other: Conventional Physical Therapy Program — The Conventional Physical Therapy Program includes the following:
  - Indoor open environment gait training exercises (over-ground gait training exercises.). (using obstacles, cones, stepper, balance board , and uneven surfaces) (either between or outside the parallel bar)
  Arms: Control Group

SUMMARY:
Safe walking needs the older adult to anticipate and respond quickly to external demands and sudden environmental changes. The practice of complex and challenging situations of the usual daily walking is very important to prevent balance loss and falls in the elderly.

Researchers reported that subjects trained in a virtual environment with enhanced feedback performed walking skills better than those trained with conventional methods. The C-Mill treadmill is an innovative device that was recently used for the training of impaired gait and balance. C-Mill treadmill uses virtual reality, augmented feedback, and force plate technology that provides the best solution for efficient functional movement therapy. Therefore, this study will evaluate the efficacy of gait training with a virtual reality treadmill on walking abilities in elderly people.

DETAILED DESCRIPTION:
Many studies have shown that walking exercises effectively contribute to enhancing walking performance in the elderly. Several studies have shown that treadmill training is effective in improving the elderly person's ability to walk. Therefore, the practice of complex and challenging situations of the usual daily walking is very important to improve walking. Unfortunately, older adults have few opportunities to practice safe walking well and consistently in a task-specific manner.

There are many studies that have shown that gait training in a challenging environment, such as walking on a treadmill, is more effective in improving the elderly person's ability to walk properly, compared to the traditional training exercise regimen that relies on training in closed training environment free from challenges and obstacles.

Virtual reality technology is one of the advanced technologies used in physical therapy and rehabilitation. This technology contributes to creating an interactive environment for the trainees that enables them to integrate into the training process and encourages them to perform controlled motor tasks. C-Mill treadmill applies a virtual reality environment, dual-tasking exercises, obstacle avoidance games, and a variety of gait challenges in a safe and controlled environment to increase walking adaptability and improve performance in everyday life. Many studies found that the C-Mill treadmill is effective in improving gait performance and adaptability in clinical practice Therefore, this study will compare the efficacy of gait training with a virtual reality treadmill and the conventional physical therapy program on walking abilities in elderly people.

ELIGIBILITY:
Inclusion Criteria:

40 healthy older adults, both sexes, will participate in this study. Their ages will be between 65 to 75 years. They should have stable medical status based on a confirmed written medical report signed by their physicians. All participants should not receive other training to improve their balance and gait during the duration of the study application except through this study training program.

Exclusion Criteria:

The exclusion criteria will include any participant with:

* a cognitive reduction (< 23 points based on the Mini-Mental State Examination scale;
* muscle paralysis,
* ﬁxed lower limb bony deformities,
* balance deficits,
* visual problems,
* diabetes mellitus,
* polyneuropathy,
* gait disorders,
* using assistive walking devices during walking,
* vertigo, anti-seizures drug use and hypertension,
* vestibular and cerebellar problems; and
* auditory and perceptual diseases/impairments

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Change in the gait parameter (stride length) (This parameter indicated the change of gait performance). | Data will be collected at baseline, 4 weeks after intervention commencement, and 4 weeks later, as follow up, after finishing the treatment program.
  An electronic walkway that connected to a portable computer will be used to measure the following gait parameter: stride length (m).
Change in the gait parameter (stride time) (This parameter indicated the change of gait performance). | Data will be collected at baseline, 4 weeks after intervention commencement, and 4 weeks later, as follow up, after finishing the treatment program.
  An electronic walkway that connected to a portable computer will be used to measure the following gait parameter: stride time (second).
Change in the gait parameter (cadence) (This parameter indicated the change of gait performance). | Data will be collected at baseline, 4 weeks after intervention commencement, and 4 weeks later, as follow up, after finishing the treatment program.
  An electronic walkway that connected to a portable computer will be used to measure the following gait parameter: cadence (steps/ minute).
Change in the gait parameter (velocity) (This parameter indicated the change of gait performance). | Data will be collected at baseline, 4 weeks after intervention commencement, and 4 weeks later, as follow up, after finishing the treatment program.
  An electronic walkway that connected to a portable computer will be used to measure the following gait parameter: velocity (meter / second).
The change in the six-minute walk test score ((This parameter indicated the change of walking tolerance abilities). | Data will be collected at baseline, 4 weeks after intervention commencement, and 4 weeks later, as follow up, after finishing the treatment program.
  The six-minute walk test (6MWT) will assess the distance that the participant's ability to walk for a total of six minutes on a hard, uneven surface. It is has been used to determine exercise tolerance changes following interventions for healthy older adults.

SECONDARY OUTCOMES:
Change in the Overall Stability Index {percentage value (%)}, and Time of Control {seconds} for Limit of Stability Test (test that assess the change in balance ability) | Data will be collected at baseline, 4 weeks after intervention commencement, and 4 weeks later, as follow up, after finishing the treatment program.
  The Biodex Balance System will be used to assess the Change in the Overall Stability Indices of the Postural Stability Test. The test includes measurement of the following indices: overall stability index, anteroposterior index and mediolateral index which represents the children's ability to control their postural balance stability in all directions. High values % represent less stability and the children had difficulty in balance control. On the other hand lower values were indicative of a better balance control.

CONTACTS AND LOCATIONS:
Overall Officials: Ehab M Abd El Kafy, PhD, Principal Investigator — Department of Physical Therapy- Faculty of Applied Medical Sciences - Umm Al Qura University
Locations (1):
- Ehab Mohamed Abd El Kafy, Mecca, Mecca Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
- The data available is Case-by-case basis at the discretion of the Primary Sponsor
Supporting Information: SAP
Time Frame: Start Date: Beginning one year following main results publication End Date: Ending two years following main results publication
Access Criteria: Data can be obtained by the Principal Investigator. Email Address: emkafy@uqu.edu.sa